## New Mexico Cancer Care Alliance University of New Mexico Cancer Center





# PROTOCOL PROTOCOL NUMBER: INST 1211

# A Pilot Randomized, Placebo Controlled, Double Blind Study of Omega-3 Fatty Acids to Prevent Paclitaxel Associated Acute Pain Syndrome

Principal Investigators: Zoneddy Dayao, MD

University of New Mexico Cancer Center 1201 Camino de Salud NE, MSC07 4025

Albuquerque, NM 87131-001

(505) 272-5490 FAX: (505) 272-7799 zdayao@salud.unm.edu

Debra Barton, RN, PhD, AOCN, FAAN

Mayo Clinic

200 First Street S.W. Rochester, MN 55905 (507) 255-3812 FAX (507) 538-8300 barton.debra@mayo.edu

Co-Investigator(s): Melanie Royce, MD

University of New Mexico Cancer Center 1201 Camino de Salud NE, MSC07 4025

Albuquerque, NM 87131-001

(505) 925-0405

FAX: (505) 272-7799 mroyce@salud.unm.edu

**Study Sites:** New Mexico Cancer Care Alliance:

University of New Mexico, Lovelace Health Systems, Presbyterian Healthcare Services, Memorial Medical Center, Christus St. Vincent Regional Medical Center, Hematology-Oncology Associates, New Mexico Cancer

Care Associates

**Study Agent:** Omega-3 Fatty Acids

Funding Source(s): NCCTG

Protocol Date:August 21, 2012; Version 1.0Revised Protocol Date:October 17, 2012; Version 2.0Revised Protocol Date:January 09, 2013; Version 3.0

April 1, 2016; Version 4.0

.

# New Mexico Cancer Care Alliance University of New Mexico Cancer Center





## **INST 1211**

#### **SIGNATURE PAGE**

The signature below constitutes the approval of this protocol and all attachments as necessary. It provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations and ICH guidelines.

| <b>Principal Inves</b> | tigator (PI) Name: Zoneddy Dayao, M.D |
|------------------------|---------------------------------------|
| PI Signature: | |
| Date: | |

#### **Background and Rationale (including feasibility)**

Paclitaxel, a widely used chemotherapeutic agent, is associated with several well-known side effects including neuropathy and generalized body aches (1). The latter has recently been described as paclitaxel- associated acute pain syndrome (P-APS) and often occurs in the 1<sup>st</sup> 3-4 days after administration (2). It affects about 58-90% of patients (2, 10). Previously, these symptoms have been described as myalgias and arthralgias (1). However, recent data support that P-APS may in fact be an early manifestation of neuropathy, as opposed to being musculoskeletal in origin. For instance, it was noted that patients with higher P-APS pain scores with the first dose of paclitaxel are at risk for developing chronic neuropathy (2, 3).

P-APS can be severe, and may require use of potent analgesics for symptom control. Non-steroidal antiinflammatory drugs (NSAIDs) are frequently used as frontline therapy. However, there is concern over side effects including gastrointestinal bleeding and acute renal injury. Many therapies have been studied including steroids (4), glutamine (5), antihistamine (6), opioid analgesics, and herbs (7), with variable results.

Low dose oral prednisone starting 24 hours after completion of chemotherapy and continued for a total of 5 days has been previously reported to result in substantial improvement in symptomatology (3). However, this study was limited due to the small sample size. In addition, given the variable schedule of paclitaxel ranging from weekly to every 3 weeks, this regimen could result in a significant amount of prednisone and can increase the risk of side effects over time.

In a placebo-controlled, double blind randomized crossover trial, the effect of glutamine on paclitaxel associated myalgias and arthralgias showed that glutamine, although well tolerated, had no effect on the development and severity of symptoms, as reported by the treating physician and by patient log (5).

Oral low-dose antihistamine, in the form of terfenadine 60 mg at the onset of pain and subsequently, has been reported to be temporarily effective in controlling paclitaxel-induced myalgia and /or dysesthesia (5). However, this study was also limited by its sample size with only 9 patients included.

Currently, there is no standard of care for P-APS. Since paclitaxel is a commonly used chemotherapeutic agent and P-APS is common and can be debilitating to some patients, an agent with a favorable toxicity profile that may prevent P-APS and possibly prevent the development of neuropathy will have significant clinical utility.

#### Data on the Pathophysiology of Paclitaxel-Associated Acute Pain Syndrome

The mechanism of P-APS is currently unknown. For many years, these subacute aches and pains were described as myalgias/ arthralgias based on patient reported symptoms. The self-limited course led to a hypothesis that symptoms are possibly the result of an inflammatory reaction to paclitaxel (1,3). More recently, Loprinzi et al reported the natural history of P-APS (2,3). In this study, P-APS symptoms were assessed in 94 patients using patients' daily symptom log with 10 items assessing pain symptoms and used of pain medication, adapted from Cleeland's Brief Pain Inventory (Appendix I). In addition, a 22-item summary questionnaire regarding symptom characteristics was given after paclitaxel use. Chemotherapy-induced peripheral neuropathy (CIPN) symptoms were assessed using the validated EORTC (European Organization for Research and Treatment of Cancer) Quality of Life Questionnaire (QLQ)-CIPN-20 given at baseline and weekly after each paclitaxel dose.

With regards to the P-APS, it was noted that the most common manifestation was a diffuse achiness mainly involving the legs, hips and lower back, typically evolving over 1-4 days. Interestingly, in the weekly paclitaxel treatment group, the initial pain experienced with the first treatment did not predict the severity of pain with additional doses, but appeared to predict the severity of symptoms associated with peripheral neuropathy, predominantly sensory, which evolved over the 12-week period of treatment. This is the first study showing that the P-APS may in fact be an early manifestation of neuropathy and is associated with the development of chronic neuropathy (2, 3).

One mechanism proposed for P-APS is an early inflammatory process characterized by macrophage activation in both the DRG and peripheral nerve occurring shortly after paclitaxel therapy (9). Morphologic alterations in DRG satellite cells have been noted and upregulation of proinflammatory cytokines have been hypothesized as early events in the development of neuropathy (9). Therefore, it is possible that paclitaxel-induced neuropathic pain may be mediated by proinflammatory cytokines. If P-APS and chronic neuropathy are indeed part of a continuum, the inflammatory pathway would be a reasonable target for therapy.

The exact mechanism on how paclitaxel eventually leads to the development of neuropathy is still not understood. Taxanes promote stabilization of microtubules leading to disruption of normal cell division, and eventually resulting in cell death. Results of a study showed that short-term administration of paclitaxel induces mainly reversible changes in the peripheral nerves and spinal roots (8). Microtubules seem to be the main target of paclitaxel neurotoxicity, in much the same way as has been described for its antineoplastic activity. It has been hypothesized that microtubule-dependent axonal transport is disrupted by paclitaxel. Abnormal aggregation of microtubules in neuronal cells is hypothesized to contribute to neurosensory abnormalities leading to impairment of axonal transport (8).

Taken together, an intervention with both anti-inflammatory as well as neuroprotective properties would be an ideal candidate for testing in the prevention of P-APS and subsequent development of peripheral neuropathy.

## Rationale for Studying Omega 3 Fatty Acids to Prevent or Ameliorate P-APS

#### Omega 3 Fatty Acids: Anti-Inflammatory Properties and P-APS.

Essential polyunsaturated fatty acids (PUFA) have two major families, the omega-6 (n-6) and omega-3 (n-3). The 20 carbon (n-3) and (n-6) fatty acids compete for the same enzymes and therefore, the intake of one omega fatty acid will diminish the metabolism of the other (10,15).

Arachidonic Acid (AA) is a primarily diet-derived 20 carbon omega-6 PUFA which serves as a precursor of proinflammatory metabolites such as prostaglandins, thromboxanes and leukotrienes (10). These eicosanoids are involved in modulating the intensity and duration of an inflammatory response. Cyclooxygenase (COX) enzymes are the rate limiting enzymes in the conversion of AA to prostaglandin E2 (PGE2) and are a target for therapy, of which the most widely studied are the NSAIDS.

Long chain omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), are common dietary supplements. They have well established anti-inflammatory properties which serve as the basis for their use in therapeutic trials in inflammatory conditions (10, 11).

EPA competes with AA for enzymatic metabolism, thereby decreasing inflammatory derivatives.

Recently, omega-3 PUFAs have also been identified as precursors of anti-inflammatory mediators called protectins and resolvins. Resolvins occur in the resolution phase of inflammation. Protectin D1 was

initially found to decrease damage of brain ischemia-reperfusion injury and thus named neuroprotectin D1 (12-14).

Several clinical studies have reported the pain relieving effects of omega 3 fatty acids for inflammatory joint diseases. In a recent meta-analysis of 17 trials, supplementation of omega-3 fatty acids for 3-4 months resulted in reduction in patient reported pain severity, duration of morning stiffness and amount of NSAID consumption (11).

As noted above, there is evidence that early inflammatory processes are observed in paclitaxel induced nerve damage. This may in part account for the symptoms of P-APS, and sustained inflammation may lead to downstream effects responsible for evolution of peripheral neuropathy (8, 9). Omega-3 fatty acids consumption can attenuate the production of pro-inflammatory metabolites. In addition, it can generate local mediators that facilitate resolution of inflammation (12-14). Thus, if P-APS is indeed mediated by inflammation, the anti-inflammatory activity of omega-3 fatty acids may be one mechanism to prevent P-APS. Additionally, given its well established safety profile, it may be an attractive alternative to NSAIDS.

### Omega 3 Fatty Acids: A Dietary Supplement with Neuroprotective Properties

The nervous system is richly endowed with omega-3 fatty acids, primarily DHA. Omega-3 fatty acids may act as natural neuroprotective agents, as well as key components in nerve hemostasis. Several studies have reported the role of omega-3 fatty acids in maintaining nerve integrity and function (16, 21). Long chain n-3 PUFAs such as docosahexaenoic acid (DHA) have been shown to have promising in the treatment of a broad range of neurodegenerative conditions (16).

Several preclinical models have shown the neuroprotective effect of DHA in models of spinal cord injury (17-19). A mouse model has recently been used comparing groups with different fatty acid profiles (19). One group expressed the *fat-1 gene* from Caenorhabditis elegans, which encodes a fatty acid desaturase, the enzyme that converts n-6 into n-3 PUFAs, leading to enrichment in tissue n-3 PUFA levels (low n-6/n-3 ratio). This was compared to the group that had a high n-6/n-3 ratio as well as to wild type strain. Utilizing in vitro and in vivo injury models, neurite growth, axonal regeneration, sensory and motor function were assessed and compared. Interestingly, the dorsal root ganglion neurons from fat-1 mice (n-3 enriched) had significant increase in neurite outgrowth and improved neuronal survival after injury. The omega-3 enriched group did not exhibit an increase in neuronal cell death after mechanical or hypoxic injury, in contrast to the 2 groups where hypoxia resulted in neuronal cell death in the order of 2.3 - 2.6 fold increase. The mice expressing the fat-1 gene showed a more complex neurite outgrowth phenotype, with neurons displaying both longer neurites and branches, supporting the notion that n-3 PUFA level had improved neuroregenerative potential. Interestingly, the in vivo experiments also showed that the higher tissue n-3 PUFA group also exhibited a faster recovery of sensory loss, as assessed by mechanical stimulation thresholds. Even after a severe form of injury such as a crush injury, recovery of sensation was faster in the group that was enriched for omega-3.

In the clinical setting, omega-3 fatty acids have been studied in a wide spectrum of neurodegenerative disorders (21- 24). Alzheimer's disease, a progressive neurodegenerative disease, has been reported to strongly correlate with decreases in omega -3 fatty acid levels in the brain and peripheral tissue compared to age-related controls (22). Epidemiological studies have also shown a correlation between lower levels of dietary omega-3 fatty acids and the development of Alzheimer's disease (23), suggesting a

neuroprotective effect. Similar observations have been seen in Parkinson's disease, a neurodegenerative disorder of the basal ganglia (24). Dietary interventions however have shown conflicting results.

There are also emerging data on the role of omega-3 fatty acid supplementation in acute neurologic injuries. As an example, it was reported that administration of moderate to high dose human albumin rich in DHA is neuroprotective in focal brain ischemia (25).

These observations lend credence to the notion that omega-3 fatty acids promote neuroprotection and neuroregeneration. These, along with its anti-inflammatory properties make it an attractive agent to study in the prevention and amelioration of paclitaxel induced peripheral neuropathy. We hypothesize that omega-3 fatty acid supplementation started prior to initiation and administration of chemotherapy can potentially attenuate paclitaxel induced nerve damage.

#### **Omega 3 Fatty Acids and Paclitaxel**

Currently, there are no documented safety concerns with the combination of omega-3 fatty acids and paclitaxel. On the contrary, preclinical and clinical studies have investigated the potential synergy with the combination treatment (26-28). In early preclinical data, sequential exposure to Omega-3 PUFA docosahexanoic acid (DHA) followed by paclitaxel or docetaxel was demonstrated to enhance cytotoxicity of taxanes against the metastatic breast cancer cell line MDA-MB-231 (26). The investigational drug Taxoprexin (DHA-Paclitaxel), a 2'-O-acyl conjugate of paclitaxel covalently bound to DHA via an ester bond, was developed to improve paclitaxel's therapeutic performance. Phase I trials did not show any dose limiting toxicities with the conjugated preparation (27). Oral omega-3 fatty acids, classified as a nutritional additive, have several commercial preparations available for over the counter use. To date, there are no reported adverse drug reactions with FDA approved Lovaza and paclitaxel.

#### **Feasibility**

P-APS is common and occurs in about 50-90% of patients. Paclitaxel is a common chemotherapeutic agent used in a variety of malignancies, both in the early and advanced setting. Therefore, it is expected that the many patients will be eligible for this clinical trial.

Omega-3 fatty acids have a well-established safety profile and have led to their wide availability and over the counter use. As detailed above, its anti-inflammatory properties and favorable side effect profile make them an attractive alternative to NSAIDS. Furthermore, its potential neuroprotective properties make them an intriguing candidate for testing in paclitaxel induced neuropathy.

This will be a multi-institutional study and the Principal Investigators are Zoneddy Dayao, MD (NCCTG) from the University of New Mexico Cancer Center and Debra Barton, RN, PhD (NCCTG) from the Mayo Clinic, Rochester, MN. Melanie Royce, MD, PhD (ACOSOG) from the University of New Mexico is a co-investigator. The primary site will be the New Mexico Cancer Care Alliance (NMCCA), as defined below.

New Mexico Cancer Care Alliance is a New Mexico nonprofit corporation established in February, 2002, that functions as a single point of contact for the management of oncology trials at multiple sites. NMCCA includes: University of New Mexico Cancer Research and Treatment Center; Lovelace Health Systems; the New Mexico Veterans Affairs Health Care System; Presbyterian Healthcare Services (Presbyterian Hospital, Presbyterian Kaseman Hospital, Presbyterian Medical Group); Memorial Medical Center, Christus St. Vincent Regional Medical Center; Hematology-Oncology Associates; New Mexico

Cancer Care Associates and New Mexico Ear, Nose, Throat Specialists, P.C.; PMG Surgery. It is a joint venture representing approximately 100 physicians in central, northern and southern New Mexico who are engaged in the care of cancer patients.

The NMCCA utilizes a centralized IRB for all participating sites: either the University of New Mexico Human Research Review Committee (HRRC), or the Western IRB. Each trial has only one full review regardless of how many sites will participate.

NMCCA has a strong commitment to clinical trial accruals. From 2010-2011, a total of 517 patients were enrolled in therapeutic and cancer control trials, with 229 from UNM and 288 from the other sites. The last 5 years have shown a steady increase in clinical trial enrollment, with a total of 2214 patients accrued at all sites from 2006-2011.

#### **B.** Aims

#### **Primary**

1. To determine whether omega-3 fatty acids can prevent or ameliorate paclitaxel associated pain syndrome (P-APS) in cancer patients.

#### **Secondary**

- 1. To determine whether omega-3 fatty acids can prevent development of peripheral neuropathy.
- 2. To assess tolerability of omega-3 fatty acids in this setting.
- 3. To compare QOL with omega-3 fatty acids supplementation versus placebo.

#### C. Study Plan

#### Eligibility criteria:

- 1. Patients have a diagnosis of breast cancer or ovarian cancer.
- 2. Patients must be  $\geq$  18 years old
- 3. Patients may be either male or female
- 4. Patients are scheduled to receive weekly paclitaxel at 70-90 mg/m2 for a minimum of 2 months. 3 out of 4 weeks is allowed.
- 5. ECOG Performance Status (PS) of 0, 1 or 2
- 6. Patients must not have taken omega-3 fatty acid supplements within the past 1 month prior to registration and must agree to refrain from use of omega-3 fatty acid supplements from sources outside the study.
- 7. Patients must not be on NSAIDS or aspirin for at least 1 week prior to registration. NSAIDS or aspirin are allowed after enrollment.
- 8. Patients must not have received any other analgesics (opiates and tramadol) 1 week prior to registration. Analgesics (opiates and tramadol) are allowed after enrollment.
- 9. Patients must have the ability to complete questionnaires by themselves or with assistance.

- 10. Patients must not be on anticoagulation medication (heparin/warfarin) within 28 days prior to registration, because of increased risk of bleeding.
- 11. Concurrent treatment with carboplatin +/- bevacizumab is allowed.
- 12. Concurrent treatment with Her2 neu targeted therapy is allowed.

#### **Exclusion Criteria**

- 1. Known allergy to omega-3 fatty acids, fish, or shellfish
- 2. Pre-existing diagnosis of peripheral neuropathy
- 3. Diagnosis of fibromyalgia
- 4. Concurrent planned neutrophil colony stimulating factor therapy
- 5. Prior exposure to paclitaxel within the last 6 months

## **Protocol Treatment:**

**Treatment:** Omega-3 Fatty Acid: 4 capsules (1 gram/capsule) or a double-blinded placebo either once daily or 2 capsules two times daily beginning 1 week prior to starting paclitaxel and continued until 12 weeks or until paclitaxel is discontinued, whichever comes first (maximum of 12 weeks).

**Rationale for dosing**: A dose of at least 2.7 g/day of EPA and DHA have been reported to have analgesic effects in inflammatory conditions (11). The dose of 4 g/day is an FDA approved dose of omega-3 fatty acids (Lovaza) for the treatment of hypertriglyceridemia and has a well-documented toxicity profile. On the basis of this, a dose of 4 g/day was selected.

**Formulation of omega-3-fatty acid:** Lovaza (omega-3-acid ethyl esters) capsules will be used. Each 1-gram capsule of Lovaza contains approximately 465 mg <u>EPA</u> and 375 mg <u>DHA</u>.

**Formulation of placebo:** Placebo will be provided by Clinical Encapsulation Services or UNM Pharmacy. Excipient material will be microcrystalline cellulose. It will be odorless like Lovaza. Since the placebo may slightly differ from Lovaza, the pills will be dispensed in opaque bottles and providers will not be allowed to open them. In addition, to document blinding, the patients will be asked on cycle 1 Day 2, if they know what medication they are receiving.

**Randomization:** Clinical Encapsulation Services or UNM Pharmacy will package both placebo and active drugs. Our pharmacy will take care of randomization. Then our research nurses will dispense the drug.

## **Measurement tools:**

**For P-APS symptoms**, there will be 4 types of questionnaires, adapted from NCCTG N08C1: (1) a baseline/pretreatment questionnaire. (2) a daily paclitaxel induced acute pain syndrome symptom log from Day 2-7 (2, 20). (3) day 8 P-APS symptom summary. (4) 1 month after completion of paclitaxel questionnaire.

**For chemotherapy-induced peripheral neuropathy (CIPN) neurotoxicity**, the EORTC-QLQ CIPN20 patient questionnaire will be used. The questionnaire will be filled out on the 8<sup>th</sup> day of each chemotherapy treatment and 1 month after completion of therapy.

**Dietary counseling**: As omega-3 fatty acid metabolism is affected negatively by the amount of arachidonic acid in the diet, dietary counseling will be provided to assess the fatty acid intake. Omega-3 and Omega-6 Fatty Acid Dietary Intake Questionnaire will be given at baseline, Week 2, Week 4 and monthly thereafter (prepared by Laura Taber, PhD).

**Laboratory tests**: Due to a small risk of increased LDL and transaminase levels, LDL and transaminase levels will be determined at baseline, at Week 4 and the last day of paclitaxel treatment.

#### **D.** Adverse Events

Adverse events (AEs) will be assessed according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.0. Adverse events will be assessed to determine tolerability as part of the secondary objectives of the study. Analyses will be performed for all patients having received at least one dose of omega-3 (Lovaza). Recording of AEs and their attribution (whether they are due to omega-3 or due to standard of care chemotherapy treatment (paclitaxel) is important to determining the tolerability of omega-3. Since this study focuses on determining whether omega-3 can prevent P-APS and/or peripheral neuropathy as well as the tolerability of omega-3 in patients undergoing treatment with paclitaxel, the scope of AE collection will be limited to:

- 1) Any AEs involving aches or pain
- 2) Any AEs involving neuropathy
- 3) Any AEs that are definitely, probably, or possibly related to omega-3/placebo or paclitaxel

In addition to recording AEs, data will be captured on whether AEs attributed to omega-3 or AEs involving aches, pains, or neuropathy cause a given patient to discontinue participation in the study. Reported adverse reactions for omega-3 fatty acids are minimal. While none of these symptoms require dose modification or discontinuation for safety concerns, patients may discontinue therapy should they choose, or if they are experiencing significant discomfort. The common side effects reported in at least 3% or greater rate than placebo in prior clinical trials using Lovaza are as follows:

- (1) Eructation (belching) which occurs in about 4%
- (2) Dyspepsia occurring in about 3%
- (3) Altered taste in about 4%
- (4) As Lovaza contains omega-3 fatty acids obtained from several fish sources, patients with known hypersensitivity or allergy to fish/shellfish are excluded. However, a person who develops a rash on the 1<sup>st</sup> week of Lovaza treatment, prior to paclitaxel administration, should be evaluated for Lovaza allergy. The rash should be graded per NCI-CTAE version 4 criteria and be recorded as a possible Lovaza allergy.

Paclitaxel Side Effects: These should be reported per NCI-CTAE version 4. Dose modification of paclitaxel will be at the discretion of the treating physician.

Side effects of paclitaxel include:

- 1) neutropenia,
- 2) transaminitis,
- 3) neuropathy,
- 4) hypersensitivity reactions,
- 5) alopecia,
- 6) arthralgias
- 7) myalgias.

Patients who discontinue paclitaxel treatment due to allergy to paclitaxel will not be evaluable.

## E. Data Analysis

In this pilot study, the effect of omega-3 on severity of paclitaxel associated pain syndrome will be evaluated in 60 patients using 1:1 randomization into omega-3 plus paclitaxel group and placebo plus paclitaxel group to achieve the primary aim. The primary endpoint will be determined by questions in N08C1 pain inventory. Mean severity will be calculated for each group and differences between groups will analyzed via t-tests or Wilcoxon rank-sum tests as appropriate. We will also consider a binary variable for incidence (no pain versus any pain, no relief versus any relief, does not interfere versus other) to evaluate the primary aim. A formal sample size justification based on statistical hypothesis is not applicable to this pilot study. Considering 60%-80% incidence of paclitaxel associated pain syndrome, we can detect a minimal difference of 37.6%-37.9% pain syndrome difference base on 5% significance level and 80% power with our proposed sample size. In this effect size calculation, the significance level actually achieved by this design is 2.2%-2.6%. Our sample size justification is based on primary aim with a binary variable of incidence.

Similarly, we will consider both continuous variables and binary incidence variable for the secondary aims. For continuous variables, t-tests or Wilcoxon rank-sum tests will be used. Fisher's exact test will be used for the incidence variable with 95% confidence intervals.

Patients will be evaluable regardless of the number of cycles of paclitaxel completed. A patient will be considered evaluable if they have completed a baseline pre-paclitaxel questionnaire and at least one questionnaire during paclitaxel treatment.

The study will last for approximately 5 years including data analysis.

### F. Data Safety Monitoring:

Data Safety Monitoring will be done by the University of New Mexico Data Safety Monitoring Board.

## G. Budget: See attached

#### H. References

1. Garrison JA, McCune JS, Livingston RB, Linden HM, Gralow JR, Ellis GK, West HL:, Myalgias and arthralgias associated with paclitaxel. Oncology 12: 271-277, 2003

- Loprinzi CL, Reeves BN, Dakhil SR, Sloan JA, Wolf SL, Burger KN, Kamal A, Le-Lindqwister NA, Soori GS, Jaslowski AJ, Novotny PJ, Lachance DH. Natural history of paclitaxelassociated acute pain syndrome: prospective cohort study NCCTG N08C1. JCO 29: 1472-1478, 2011
- 3. Reeves, Dakhil et al: Further data supporting that paclitaxel-associated acute pain syndrome is associated with development of peripheral neuropathy. Cancer, 2012
- 4. Markman M, Kennedy A, Webster K, Kulp B, Peterson G, Belinson J. Use of low dose oral prednisone to prevent paclitaxel- induced arthralgias and myalgias. Gynecol Oncol Jan 72 (1) 100-101, 1999
- Jacobson SD, Loprinzi CL, Sloan JA, Wilke JL, Novotny PJ, Okuno SH, Jatoi A, Moynihan TJ Glutamine does not prevent paclitaxel- associated myalgias and arthralgias. The Journal of Supportive Oncology; 1:274-278, 2003
- 6. Martoni A, Zamagni C, Gheka A, Pannuti F Antihistamines in the treatment of taxol-induced paroxystic pain syndrome. J Natl Cancer Inst 85;676, 1993
- 7. Yoshido T, Sawa T, Ishiguro T, Horiba A, Minatoguchi S, Fujiwara H. The efficacy of prophylactic shakuyaku-kanzo-to for myalgia and arthralgia following carboplatin and paclitaxel combination chemotherapy for non-small cell lung cancer. Support Care Cancer Mar 17(3):315-20, 2009.
- 8. Peters CM, Jimenez-Andrade JM, Jonas BM, Secik MA, Koewler NJ, Ghilardi JR, Wong GY, Mantyh PW. Intravenous paclitaxel administration in the rat induces a peripheral sensory neuropathy characterized by macrophage infiltration and injury to sensory neurons and their supporting cells. ExpNeurol Jan; 203 (1), 2007
- 9. Cavaletti G, Cavalleti E, Montaguti P, Oggioni N, De Negri O, Tredici G. Effect on the peripheral nervous system of the short-term intravenous administration of paclitaxel in the rat. Neurotoxicology 18 (1): 137-45, 1997
- 10. Calder PC. Polyunsaturated fatty acids, inflammatory processes and inflammatory bowel diseases. Mol Nutr Food Res 52; 885-97, 2008
- 11. Goldberg, RJ, Katz, J. A meta-analysis of the analgesic effects of omega-3 polyunsaturated fatty acid supplementation for inflammatory joint pain. Pain 129 210-223, 2007
- 12. Hong S. Gronert K Serhan C. Novel docosatrienes and 17S-resolvins generated from docosahexaenoic acid in murine brain, human blood, and glial cells. Autacoids in anti-inflammation. J Biol Chem 278 (17): 14677-97, 2003
- Marcheselli VL, Hong S, Lukiw Wj et al. Novel docosanoids inhibit brain ischemia-reperfusionmediated leukocyte infiltration and pro-inflammatory gene expression. J Biol Chem 278 (44): 43807-17, 2003
- 14. Ru-Rong Ji Emerging Roles of Resolvins in the resolution of inflammation and pain. Trends in Neurosciences, November Vol. 34, No 11, 2011
- 15. Whelan J, McEntee MF Dietary (n-6) PUFA and intestinal tumorigenesis J Nutr Dec; 134 (12 Suppl) 3421S-3426S, 2004

- 16. Bazan, N. Docosahexaenoic acid signalolipidomics in nutrition: significance in aging, neuroinflammation, macular degeneration, alzheimer's, and other neurodegenerative diseases. Annu. Rev. Nutr. 31:321-51, 2011
- 17. King VR, Huang WL, Dvall SC, Curran OE, Priestley JV, Michell-Titus AT. Omega 3 fatty acids improve recovery, whereas omega 6 fatty acids worsen outcome, after spinal cord injury in the adult rat. J Neurosci. April 26; 26(17) 4672-80, 2006
- Lim SN, Huang W, Hall JC, Ward RE, Priestley JV, Michell- Titus AT. The acute administration of eicosapentaenoic acid is neuroprotective after spinal cord compression injury in rats Prostaglandins Leukotr Essent Fatty Acids Oct- Dec; 83 (4-6) 193-201, 2010
- 19. Gladman S, Huang W, Lim, S, Dyall S, Boddy, S, Kang, J, Knight, M, Priestley J, Michael-Titus AT. Improved outcome after peripheral nerve injury in mice with increased levels of endogenous omega-3 polyunsaturated fatty acids The Journal of Neuroscience January 11 32(2): 563-571, 2012
- 20. Cleeland C: How to assess cancer pain, in Tuck DC, Medzak R (eds): Handbook of Pain Assessment. New York, NY. The Guilford Press, pp 360-387, 1992
- 21. Dyall, SC., Michael-Titus AT. Neurological Benefits of Omega-3 Fatty Acids. Neuromol Med 10:219-235, 2008
- 22. Kyle, DJ, Schaefer, E., Patton, G., Beiser, A. Low serum docosahexaenoic acid is a significant risk factor for Alzhemier's dementia. Lipids, 34 (Suppl) S245, 1999
- 23. Barberger-Gateau, P., Letenneur, L., Deschamps, V. Peres, K. Dartigues, JF, Renaud S. Fish, meat and risk of dementia: Cohort study. British Medical Journal, 325, 932-933, 2002
- De Lau, LM, Bornebroek, M. Witteman, JC., Hofman, A. Koudstaal, PJ, Breteler MM. Dietary fatty acids and the risk of Parkinson disease: The Rotterdam study, Neurology, 64 (12), 2040-2045, 2005
- 25. Belyev, L, Liu Y. Zhao W, Busto R, Ginsberg, MD Human albumin therapy of acute ischemic stroke: Marked neuroprotective efficacy at moderate doses and with a broad therapeutic window. Stroke 32(2), 553-560, 2001
- 26. Menendez JA, Lupu R, Colomer R. Exogenous supplementation with omega -3 polyunstaurated fatty acid docosahexanoic acid (DHA; 22: 6n3) synergistically enhances taxane cytotoxicity and downregulates Her2/neu (c-erbB-2) oncogene expression in human breast cancer cells: Eur J Cancer Prev Jun;14 (3) 263-70, 2005
- 27. Fracasso PM, Picus J, Wildi JD, Goodner SA, Creekmore AN, Gao F, Govindan R, Ellis MJ, Tan BR, Linette GP, Fu CJ, Pentikis HS, Zumbrun SC, Egorin MJ, Bellet RE. Phase 1 and Pharmacokinetic study of weekly docosahexanoic acid-paclitaxel Taxoprexin, in resistant solid tumor malignancies: Cancer Chemother Pharmacol, Feb;63(3); 451-8, 2009

| Test and Procedures | Baseline<br>(Baseline or <28<br>days after<br>registration) | Daily, Days 2-7<br>following each<br>paclitaxel dose | Day 8 following<br>each paclitaxel<br>dose | 1 Month after<br>completion of<br>Therapy |
|---|---|---|---|---|
| Baseline Pre-<br>Paclitaxel<br>Questionnaire<br>(Appendix 1) | x | | | |
| Toxicity (AE)<br>Assessment | x | | X<br>(+/- 3 days) | Х |
| Daily Paclitaxel-<br>Induced acute pain<br>Syndrome Symptom<br>Log (Appendix II) | | X **On Day 2 of cycle 1 only, patients will answer question #11 | | |
| Day 8 PAPS Symptom<br>Summary<br>Questionnaire<br>(Appendix III) | | | х | |
| EORTC QLQ-CIPN20<br>Questionnaire<br>(Appendix IV) | | | х | x |
| 1 Month post<br>paclitaxel<br>Questionnaire<br>(Appendix V) | | | | x |
| Dietary Counseling | X | | | |
| Dietary Questionnaire<br>(Appendix VI) | | | Week 2 and Week 4,<br>then monthly<br>thereafter | x |
| Lipid panel | x | | Week 4 | X |
| LFTs | x | | Week 3 or 4 | |

#### APPENDIX I

#### **Baseline Pre-paclitaxel Questionnaire**

| Pa | tient Study ID Num | ber: | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Da | te: | | | | | | | | | | |
| Dir | ections: Please an | swer the | following q | uestions: | | | | | | | |
| 1. | Do you have any | chronic a | aches and pa | ains? (Circle | e Yes or No | ) | | | | | |
| | Yes | | | No | | | | | | | |
| 2. | Do you regularly | take pair | n medication | ns? (Circle \ | es or No) | | | | | | |
| | Yes | | | No (If no, | go to ques | tion 4) | | | | | |
| 3. | If yes, please list t | he name | of each med | lication: | | | | | | | |
| 4 | How much of a p | oroblem v | vas numbne | ss and/or t | ingling in y | our hands ( | or fingers <u>ov</u> | ver the last | week (circle | one numb | per)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No<br>numbness or<br>tingling | | | | | | | | | | Jumbness/tingling<br>s bad as it can be |
| 5 | How much of a pro | oblem wa | s numbness | and/or tin | gling in you | ır feet or to | es <u>over the</u> | last week | (circle one i | number)? | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No numbness or tingling | | | | | | | | | | Numbness or<br>tingling as<br>bad as it can<br>be |
| 6. | . How much of a p | roblem w | as burning o | or shooting | PAIN in yo | ur hands ar | nd fingers <u>o</u> | ver the last | week (circle | e one numl | ber)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No pain | | | | | | | | | | Pain as bad as it can be |
| 7. | How much of a p | roblem w | as burning c | or shooting | PAIN in yo | ur feet or t | oes <u><b>over th</b>e</u> | e last week | (circle one | number)? | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No pain | | | | | | | | | | Pain as bad as it can be |

# Appendix II

# Daily Paclitaxel- Induced Acute Pain Syndrome Symptom Log

| v# | | Date:_ | | _ | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. | | | | | | | | | | | might be related to |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No | | | | | | | | | | Aches/pains as bad |
| | pain | | | | | | | | | | as can be |
| 2. | Please i | rate the s | ame aches | s/pains by | circling th | e ONE n | umber that | best desc | ribes your | pain at i | ts <b>LEAST in the la</b> |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No | | | | | | | | | | Aches/pains as bad |
| | pain | | | | | | | | | | as can be |
| 3. | | rate the s 24 hour | | s/pain by | | | | | | 9 | ins on the <b>AVERAC</b> 10 ches/pains as bad |
| | pain | | | | | | | | | ; | as can be |
| 4. | | | nonprescr<br>e Yes or N | | dication, li | ke aspirir | n , Tylenol | , Motrin, l | buprofen | or Advil | , for the pain in the |
| | Yes | | No (I | f no, go to | o question | 7) | | | | | |
| | | | | | medication | | | | | | |

| 6. | | | te by circli<br><b>24 hours</b> . | ing ONE 1 | number ho | w helpful | these non | prescriptio | on medica | tions we | re in controlling your |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No | | | | | | | | | | Aches/pains as bad pain as can be |
| 7. | Have y | | opioid med | lications l | like codeir | ie, oxycod | lone or mo | orphine for | this pain | in the la | st 24 hours ( Circle Yes |
| | Yes | 1 | No (If no, | go to ques | stion 10) | | | | | | |
| 8. | If yes, | please lis | st the nam | e of each | medicatio | n: | | | | | |
| | | | | _ | | | | | | _ | |
| | | | | _ | | | | | | _ | |
| 9. | | please ra | | ing ONE | number h | ow helpfu | l these opi | oid pain n | nedication | s were in | n controlling your pain in |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not he | lpful, | | | | | | | Complete | ly helpfu | ıl |
| | No pain | control | | | | | | | | No pain | after taking drug |
| 10. | Other | comment | ts: | | | | | | | | |
| 11. | Day | 2 Cycle 1 | only: | | | | | | | | |
| | What di | rug do yo | u think yo | u are taki | ng? Plac | cebo | Lovaza | I don' | t know/ I | can't tell | |

#### APPENDIX III

Day #8 Paclitaxel-induced Acute Pain Syndrome Symptom Summary

| Pat | tient Study ID Numb | oer: | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Da | te: | | | | | | | | | | |
| Dir | ections: Please ans | wer the f | ollowing que | estions: | | | | | | | |
| 1. | Over the previous | | | | NEW ache | es/pains that | you did no | ot have prio | r to your la | st dose of o | chemotherapy and |
| | Yes | | | No | | | | | | | |
| | If NO, then | you can : | skip to quest | tion 18. | | | | | | | |
| 2. | Please rate any a | ches/pai | ns that you h | nave by circ | ling <b>ONE</b> n | umber that I | oest descrik | oes your acl | nes/pains a | t its worst | over the last week |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No aches or pains | | | | | | | | | | Aches or pains as bad as can be |
| 3. | Please place a <b>CHEC</b> | к mark (v | /) by all of th | ne appropri | ate words t | that could be | e used to de | escribe this | | pain? | |
| | Sharp | | | | | | | | | | |
| | Dull | | | | | | | | | | |
| | Throbbing | | | | | | | | | | |
| | Cramping | | | | | | | | | | |
| | Stabbing | | | | | | | | | | |
| | Gnawing | | | | | | | | | | |
| | Burning-ho | t | | | | | | | | | |
| | Aching | | | | | | | | | | |
| | Heavy | | | | | | | | | | |
| | Splitting | | | | | | | | | | |
| | Shooting | | | | | | | | | | |
| | Stinging | | | | | | | | | | |
| | Pulsating | | | | | | | | | | |

| 4. | Please place a <b>CHECK</b> mark (V) by the two words that are most descriptive of your pain: |
|---|---|
| | Sharp |
| | Dull |
| | Throbbing |
| | Cramping |
| | Stabbing |
| | Gnawing |
| | Burning-hot |
| | Aching |
| | Heavy |
| | Splitting |
| | Shooting |
| | Stinging |
| | Pulsating |
| 6.<br>app | Please indicate where these <b>NEW</b> pains are/were located by placing a <b>CHECK</b> mark (v) next to the location(s), please mark all that ly: |
| | Arms, above the elbow |
| | Arms, between the elbows and wrists |
| | Hands |
| | Legs above knee |
| | Legs, between the knee and ankles |
| | Feet |
| | Upper back |
| | Lower back |
| | Neck |
| | Head |
| | Chest |

| | Abdomen | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Hips | | | | | | | | | | |
| | Shoulders | | | | | | | | | | |
| | Other, please | specify | | | | | | | | | |
| 7. | Please note wh | nether walki | ng or stand | ing increase | ed any new | pain that ye | ou had after | the paclita | ixel you red | ceived (Circl | e one number) |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all | | | | | | | | | | Yes, quite a bit |
| 8.<br>num | Please note whaber) | nether light | touching of | areas of pa | in increased | d any new p | pain that you | u had after | the paclitax | el you rece | ived. (Circle one |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all | | | | | | | | | | Yes, quite a bit |
| 10. | or no) Yes If yes, please lis | st each med | lication and | | go to questi<br>ow many yo | | each over th | e past weel | k: | | |
| | Medicatio | on: | | | | | Number us | ed over the | past week | | |
| | | | | _ | | | | | | | |
| 11. | If yes, please ra | ate by circlin | ig <b>ONE</b> num | ber how he | elpful these | nonprescri | ption medic | ations were | e in controll | ing your pa | in <u>overall during the</u> |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not helpful,<br>no pain<br>control | | | | | | | | | | Extremely<br>helpful, no<br>pain after<br>taking the<br>drug(s) |
| 12 | Have you used | d opioid pai | n medicatio | ns (e.g. cod | eine, oxyco | done, morr | ohine, etc) fo | or this pain | over the la | <u>st week</u> ? (C | ircle Yes or No) |
| | Yes | | | No (If no, | go to questi | ion 15) | | | | | |

| | Medicatio | n: | | 1 | Number use | ed over the | past week: | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 14. | If yes, please rate | te by circlir | ng <b>ONE</b> num | ber how he | lpful these | opioid pain | n medications | s were in c | ontrolling y | our pain | overall during the last |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not helpful,<br>no pain<br>control | | | | | | | | | | Extremely<br>helpful, no<br>pain after<br>taking the<br>drug(s) |
| 15 | Have you used | anything e | lse (e.g. mas | sage, whirl | pool, streto | ching, etc) fo | or this pain <u>o</u> | ver the las | st week? (C | Circle Yes o | or No) |
| | Yes | | | No | | | | | | | |
| 16. | If yes, please spe | ecify: | | | | | | | | | |
| 17. | If yes, please ra | te by circlir | ng <b>ONE</b> num | ber how he | lpful these | things were | e in controllir | ng your pa | in <b>overall o</b> | during the | last week. |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not helpful,<br>no pain<br>control | | | | | | | | | | Extremely<br>helpful, no pain<br>after taking the<br>treatment (s) |
| 18. | How much of a p | roblem wa | s numbness | and/or ting | gling in you | r hands or f | ingers <u>over t</u> | he last we | <u>eek</u> (circle d | one numb | er)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No numbness or tingling | | | | | | | | | | Numbness or<br>tingling as<br>bad as it can<br>be |

13. If yes, please list each medication and estimate how many you took of each over the past week:

| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | No numbness or tingling | | | | | | | | | | Numbness or<br>tingling as<br>bad as it can<br>be |
| 20. | How much of a pr | oblem wa | ıs burning oı | rshooting F | AIN in your | hands or fi | ngers <u>over</u> | the last we | <u>ek</u> (circle o | ne numbe | r)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No pain | | | | | | | | | | Pain as bad as<br>it can be |
| 21. | How much of a pr | oblem wa | s burning o | r shooting F | PAIN in your | feet or toe | s <u>over the l</u> | ast week | (circle one | number)? | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | No pain | | | | | | | | | | Pain as bad as it can be |

## APPENDIX IV

# EORTC QLQ- CIPN20

| Patient Study ID Number: |
|--------------------------|
|--------------------------|

Date:\_\_\_\_\_

| During the past week: | Not at all | A little | Quite a Bi | t Very much | 1 |
|---|---|---|---|---|---|
| 1. Did you have tingling fingers or hands? | | 1 | 2 | 3 | 4 |
| 2. Did you have tingling toes and feet? | | 1 | 2 | 3 | 4 |
| 3. Did you have numbness in your fingers/ hands? | | 1 | 2 | 3 | 4 |
| 4. Did you numbness in your toes or feet? | | 1 | 2 | 3 | 4 |
| 5. Did you have shooting or burning pain in your fi hands? | ngers/ | 1 | 2 | 3 | 4 |
| 6. Did you shooting or burning pain in your toes ar | nd feet? | 1 | 2 | 3 | 4 |
| 7. Did you have cramps in your hands? | | 1 | 2 | 3 | 4 |
| 8. Did you have cramps in your feet? | | 1 | 2 | 3 | 4 |
| 9. Did you have problems standing or walking bed of a difficulty feeling the ground under your feet? | cause | 1 | 2 | 3 | 4 |
| 10. Did you have difficulty distinguishing between water? | hot and cold | 1 | 2 | 3 | 4 |
| 11. Did you have a problem holding a pen, which r difficult? | made writing | 1 | 2 | 3 | 4 |
| 12. Did you have difficulty manipulating small objections your fingers (for example, fastening small buttons) | | 1 | 2 | 3 | 4 |
| 13. Did you have difficulty opening a jar or bottle of weakness in your hands? | because | 1 | 2 | 3 | 4 |
| 14. Did you difficulty walking because your feet dr downwards? | opped | 1 | 2 | 3 | 4 |
| 15. Did you have difficulty climbing stairs or gettir of a chair because of weakness in your legs? | ng up out | 1 | 2 | 3 | 4 |
| 16. Were you dizzy when standing up from a sitti lying position? | ng or | 1 | 2 | 3 | 4 |
| 17. Did you have blurred vision? | | 1 | 2 | 3 | 4 |
| 18. Did you have difficulty hearing? | | 1 | 2 | 3 | 4 |
| 19. If you drive a car, did you have difficulty using | pedals? | 1 | 2 | 3 | 4 |
| 20. (Answer only if you are a man) Did you have difficulty getting or maintaining an erection? | | 1 | 2 | 3 | 4 |

# Appendix V

# Monthly Questionnaire after paclitaxel chemotherapy completion

| Patient S | Study ID Number: | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Date: | | | | | | | | | | | | |
| 1. How | much of a prob | lem wa | s numbr | iess and, | or tingli/ | ng in yo | ur hands | or finge | ers <u>over t</u> | the last v | veek (circle one | 9 |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | No<br>numbness<br>or<br>tingling | | | | | | | | | | Numbness<br>or tingling<br>as bad as<br>it can be | |
| 2. How | much of a prob | lem wa | s numbr | ess and, | or tingli/ | ng in yo | ur feet o | r toes <u>o</u> | ver the la | ast week | (circle one nun | nber)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | No<br>numbness<br>or<br>tingling | | | | | | | | | | Numbness<br>or tingling<br>as bad as<br>it can be | |
| 3. How | much of a prob | lem wa | s burnin | g or sho | oting PA | IN in you | ır hands | or finge | rs <u><b>over t</b></u> | he last w | <u>reek</u> (circle one | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | No pain | | | | | | | | | | Pain as<br>bad as it<br>can be | |
| 4. How | much of a prob | lem wa | s burnin | g or sho | oting PA | IN in yοι | ır feet or | toes <u>ov</u> | er the la | st week | (circle one num | ıber)? |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | No pain | | | | | | | | | | Pain as bad as it can be | |
| | 6. Other Comr | nents: | | | | | | | | | | |

**APPENDIX VI** 

#### **OMEGA-3 and OMEGA-6 FATTY ACID DIETARY INTAKE QUESTIONNAIRE**

| Patient Study ID Number: |
|--------------------------|
| Date: |

<u>Instructions</u>: You will be asked to complete this form at the time of registration, and every two weeks for the first month of the study. After that, you will be asked to complete this form at the completion of the study.

By selecting one (1) box per line, please indicate your average use, during the past 2 weeks, of each specific food. Please select a box by marking an "X" in it for one serving, or two or more "X 's" for more than one serving.

3 oz = the size of a deck of cards

| | Never or less than once per | 1<br>per | 2<br>per | 3<br>per | 4<br>per | 5<br>per | 6<br>per | 7 per<br>week | 2<br>per | 3+<br>per |
|---|---|---|---|---|---|---|---|---|---|---|
| Food | week | week | week | week | week | week | week | (every<br>day) | day | day |
| Whole egg | | | | | | | | | | |
| Canned tuna fish | | | | | | | | | | |
| (3 oz) | | | | | | | | | | |
| Dark meat fish (i.e.<br>salmon, mackerel,<br>sardines, swordfish)<br>(3 oz) | | | | | | | | | | |
| White fish (3 oz) | | | | | | | | | | |
| Shrimp or lobster (3 oz) | | | | | | | | | | |
| Scallops (3 oz) | | | | | | | | | | |
| Chicken – white meat (3 oz) | | | | | | | | | | |
| Chicken – dark meat<br>(3 oz) | | | | | | | | | | |
| Turkey – white meat (3 oz) | | | | | | | | | | |
| Turkey – dark meat (3 oz) | | | | | | | | | | |

| Beef (hamburger, ribs or steak) |
|--------------------------------------|
| (3 oz) |
| Pork (pork chop, ribs, ham or roast) |
| (3 oz) |
| Pork or beef chile or stew (1/2 cup) |
| Chicken or pork posole (1/2 cup) |
| Chicken or beef taco or burrito |
| (1 medium) |

APPENDIX VII

## **Dietary Information**

Part of this study is to collect information regarding your diet since there are certain foods rich in arachidonic Acid that can lower the effects of omega-3 fatty acids.

Arachidonic Acid (omega-6) rich foods

EPA and DHA (omega-3) rich foods

Egg yolks

Chicken Shellfish

Turkey Beef

Pork

Fish

APPENDIX VIII

# **INST 1211 Questionnaire Summary Checklist:**

| Patient Name: | | | |
|---|---|---|---|
| Patient Study ID #: | | | |
| Date Range: to | | | |
| This form is a checklist for use by the research coordinator. Please us collected. After obtaining the patient's signature, please file this form | | _ | ch questionnaires are |
| Questionnaires: | | | |
| Baseline Pre-paclitaxel Questionnaire | ☐ Yes | □No | □N/A |
| Daily Paclitaxel Induced Pain Syndrome Symptom Log | ☐ Yes | □No | □N/A |
| Days 2 through 7 of Cycle | | | |
| Day 8 Paclitaxel-Induced Acute Pain Syndrome Symptom Summary | ☐ Yes | □No | □N/A |
| EORTC QLQ-CIPN20 | ☐ Yes | □No | □N/A |
| Monthly Questionnaire after Paclitaxel Chemotherapy Completion | ☐ Yes | □No | □N/A |
| Omega-3 and Omega-6 Fatty Acid Dietary Intake | ☐ Yes | □No | □N/A |
| I have completed the above documents as indicated above and have | returned them | to the clinic on t | he date below. |
| Patient Signature | Date | | |
| Study Team Member Signature | Date | | |

How this pilot study will lead to an ALLIANCE protocol

This pilot study will explore the role of omega 3 fatty acids in preventing or ameliorating the severity of paclitaxel associated acute pain syndrome (P-APS) and development of peripheral neuropathy in cancer patients. This will be a multi-institutional study conducted by the University of New Mexico under the auspices of the New Mexico Cancer Care Alliance (NMCCA), a nonprofit corporation with approximately 100 physicians in central, northern and southern New Mexico. The NMCCA functions as a single point of contact for clinical trials. Through this organization, cooperative trials including NCCTG, ACOSOG and CALGB, have been opened and several patients have been accrued.

This feasibility trial will provide an opportunity for three investigators from the legacy groups to collaborate: Zoneddy Dayao, MD (NCCTG), Debra Barton, RN, PhD (NCCTG) and Melanie Royce, MD, PhD (ACOSOG). This also provides an opportunity for mentoring a junior faculty in the conduct of symptom intervention trial. If the results are positive, a definitive ALLIANCE Phase III trial will be conducted. The legacy group NCCTG, now ALLIANCE have conducted and published the largest body of evidence in P-APS and CIPN. Well established methodologies as well as correlative studies from the NCCTG experience will be used to further enhance the design of the Phase III trial. Given the straightforward intervention schema and the high incidence of P-APS, rapid accrual to this trial is anticipated.

Other support for this project: Currently none.